CLINICAL TRIAL: NCT01377935
Title: Comparison of Risk of Hospitalization for Acute Kidney Injury Between Patients With Type 2 Diabetes Initiating Saxagliptin and Those Initiating Other Oral Antidiabetic Treatments
Brief Title: Risk of Acute Kidney Injury Among Patients With Type 2 Diabetes Exposed to Oral Antidiabetic Treatments
Status: Completed | Type: Observational
Sponsor: AstraZeneca (Industry)
Collaborators: Bristol-Myers Squibb (Industry); University of Pennsylvania (Other)
Responsible Party: Sponsor
Other Study IDs: CV181-157
Record Dates: First submitted 2011-06-20; First posted 2011-06-22 (Estimated); Last update posted 2016-09-20 (Estimated); Status verified 2016-09

CONDITIONS: Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Observational Model: Cohort
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Patients exposed to Saxagliptin
- Patients exposed to OAD in classes other than DPP4 inhibitors: OAD - Oral Antidiabetic Drug

SUMMARY:
The purpose of this study is to compare the incidence of hospitalization for acute kidney injury among patients with type 2 diabetes who are new initiators of Saxagliptin and those who are new initiators of other oral antidiabetic drugs in classes other than Dipeptidyl peptidase IV (DPP4) inhibitors.

DETAILED DESCRIPTION:
Prospectively designed retrospective database study. This study will be conducted using administrative claims data and electronic medical records that are collected as part of routine clinical practice.

This will be a prospectively-designed database cohort study comparing hospitalizations for acute kidney injury among new initiators of Saxagliptin compared to those who are new initiators of OADs in classes other than DPP4 inhibitors. The study time frame will be from 2009 through 2014.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or older
* Newly prescribed Saxagliptin or an OAD in a class other than DPP4 inhibitors
* Enrolled in the respective database for at least 180 days prior to the first prescription of new OAD

Exclusion Criteria:

* Patients identified with a diagnostic code for acute kidney injury within the 180-day baseline period
* Patients with DPP4 inhibitor exposure during the baseline period
* Patients currently using Exenatide or Insulin

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This study will carried out using databases containing administrative claims data [ HealthCore Integrated Research DatabaseSM (HIRD) and Medicare in the U.S.] and electronic medical records [ General Practice Research Database (GPRD) and The Health Improvement Network (THIN) in the UK]. The US population includes patients from health plans in the northeast, southeastern, mid-Atlantic, central, mid-western, and western regions (HIRD) as well as US citizens 65 years of age and older (Medicare). The UK population includes patients seeking medical care from general practitioners (GPRD and THIN).
Sampling Method: Non-Probability Sample
Enrollment: 113505 (Actual)
Dates: Start 2009-08; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Hospital admission for acute kidney injury | 52 months

SECONDARY OUTCOMES:
Deaths due to acute kidney injury | 18 months
Deaths due to acute kidney injury | 36 months
Deaths due to acute kidney injury | 54 months
Hospitalizations for acute kidney injury and/or death due to acute kidney injury | 18 months
Hospitalizations for acute kidney injury and/or death due to acute kidney injury | 36 months
Hospitalizations for acute kidney injury and/or death due to acute kidney injury | 54 months

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb

REFERENCES:
- [Derived] Lo Re V, Carbonari DM, Saine ME, Newcomb CW, Roy JA, Liu Q, Wu Q, Cardillo S, Haynes K, Kimmel SE, Reese PP, Margolis DJ, Apter AJ, Reddy KR, Hennessy S, Bhullar H, Gallagher AM, Esposito DB, Strom BL. Postauthorization safety study of the DPP-4 inhibitor saxagliptin: a large-scale multinational family of cohort studies of five outcomes. BMJ Open Diabetes Res Care. 2017 Jul 31;5(1):e000400. doi: 10.1136/bmjdrc-2017-000400. eCollection 2017. PMID 28878934
- [Derived] Saine ME, Carbonari DM, Newcomb CW, Nezamzadeh MS, Haynes K, Roy JA, Cardillo S, Hennessy S, Holick CN, Esposito DB, Gallagher AM, Bhullar H, Strom BL, Lo Re V 3rd. Determinants of saxagliptin use among patients with type 2 diabetes mellitus treated with oral anti-diabetic drugs. BMC Pharmacol Toxicol. 2015 Apr 2;16:8. doi: 10.1186/s40360-015-0007-z. PMID 25889498
- See also: BMS Clinical Trials Disclosure — http://www.bms.com/clinical_trials/Pages/home.aspx
- See also: Investigator Inquiry form — http://www.bms.com/clinical_trials/Pages/Investigator_Inquiry_form.aspx
- See also: For FDA Safety Alerts and Recalls refer to the following link — http://www.fda.gov/Safety/MedWatch/SafetyInformation/default.htm
- See also: CSR Synopsis — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_MED_7111&studyid=4448&filename=cv181_157.pdf